CLINICAL TRIAL: NCT04331431
Title: Professor of Neurosurgery
Brief Title: Outcomes of the Intradural Extramedullary Tumors Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, ahmed salaheldin mohammed saro, Assistant professor of neurosurgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sohag77
Record Dates: First submitted 2020-03-28; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Spinal Cord Tumor
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spinal cord tumors (Other)
  Interventions: Procedure: Spinal cord tumor resection

INTERVENTIONS:
Procedure: Spinal cord tumor resection — Excision of intradural tumors

SUMMARY:
The intradural extramedullary tumors remain curable diseases. Our aim in this study is to evaluate the postoperative status after the tumor resection and compare it to the preoperative status

DETAILED DESCRIPTION:
Meticulous microscopic excision without nerve root or dural injuries

ELIGIBILITY:
Inclusion Criteria:

* neurological deficit
* back pain

Exclusion Criteria:

* old age above 80 years
* immunocompromised patients

Ages: 28 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-08 (Actual)

PRIMARY OUTCOMES:
complete excision | 7 years
  delicate dissection